CLINICAL TRIAL: NCT05959603
Title: Intra-wound Vancomycin Powder for Prevention of Surgical Site Infection Following Spinal Surgery - a Randomized Controlled Superiority Trial
Brief Title: Intra-wound Vancomycin Powder for Prevention of Surgical Site Infection Following Spinal Surgery
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Eyal Itshayek, Prof. Eyal Itshayek, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RMC 0103-20
Record Dates: First submitted 2021-05-20; First posted 2023-07-25 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-07

CONDITIONS: Infection
Keywords: Vancomycin; Infections; Surgical Site
MeSH Terms: conditions — Infections | interventions — Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Standard of care (No Intervention): 2 g of IV cefazolin will be administered within 60 minutes before surgical incision (3 g for pts weighing ≥120 kg), repeated dose in the operating room every four hours (allergic patients will receive 900 mg of clindamycin within 60 minutes which will be repeated every six hours or 15 mg/kg of vancomycin once within two hours before incision).
- Intervention group: 500 mg vancomycin (Experimental): Patients will receive 500 mg of powdered vancomycin to the surgical site in addition to standard of care IV prophylaxis
  Interventions: Drug: Vancomycin
- Intervention group: 1 g vancomycin (Experimental): Patients will receive one gram of powdered vancomycin to the surgical site in addition to standard of care IV prophylaxis
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Vancomycin — Powdered vancomycin will be locally administered once during surgery. The vancomycin will be placed in the surgical bed at several layers: around the hardware and before muscle apposition and above the fascia. This is done before the closure of the muscular fascia and skin by the neurosurgeon. The vancomycin will not be mixed in the bone graft.
  Arms: Intervention group: 1 g vancomycin; Intervention group: 500 mg vancomycin

SUMMARY:
Cefazolin is given routinely pre and intraoperatively for patients undergoing spinal surgery to reduce the rate of infection. Intra-wound admission of Vancomycin powder has been suggested to reduce wound infection rates. Therefore, this study aims to compare the rate of wound-related complications between patients receiving standard treatment compared to patients receiving an addition of topical Vancomycin and to identify the optimal Vancomycin dosage. All groups will receive the recommended regimen of routine IV antibiotic prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing posterior spinal fusion operation at the neurosurgery department at the Rabin Medical Center
* Ability to understand and sign written informed consent by the patient or legal guardian

Exclusion Criteria:

* Preoperative ongoing infectious disease present as judged by the primary surgeon (based on lab results and clinical assessment)
* Receiving ongoing treatment of antibiotics for other infections
* Sensitivity or allergy to vancomycin or cefazolin
* Previous spine surgery at the index level within the last 90 days
* Postoperative radiotherapy of the surgical site required (e.g. for tumor)
* Renal insufficiency with stage 4 chronic kidney disease (CKD) with a glomerular filtration rate (GFR) of 15-30 ml/min or worse
* Undergoing spinal decompression only
* Trauma patients
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363 (Estimated)
Dates: Start 2020-05-31 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of deep spinal infections | One year
  According to Center for Disease Control and Prevention (CDC) criteria

SECONDARY OUTCOMES:
Incidence of superficial spinal infections | One year
  According to CDC criteria
Individual components of the composite primary outcomes | One year
  Deep surgical site infections and superficial surgical site infections separately
Rate of Surgical site infection revisions | 30 days
  Number of surgical site infection revisions
Number of adverse events | Up to one week post-surgery
  Number of adverse events Including rash, acute kidney injury (according to RIFLE criteria, see appendix), ototoxicity
Length of hospitalization | From operation date to discharge (up to 4 weeks) or date of death
  Length of hospitalization starting on operation date up to discharge or death
Rate of mortality | One year
  Rate of mortality among study participants within one year from operation date
Rate of post-operative seroma | 30 days
  Rate of post-operative seroma
Concentration of creatinine (mg/dl), glucose (mg/dl) and albumin (g/dl) | Pre-operation, Post-operation Day 3, Post-operation Day 7, Post-operation Day 30
  Creatinine, glucose and albumin lab results
Serum vancomycin levels | 6 and 12 hours post op and then one test a day until vancomycin levels reach zero
  Serum vancomycin levels

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Itshayek, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: Undecided